CLINICAL TRIAL: NCT00573404
Title: A Phase I Study of Imatinib Mesylate and SU011248 for Patients With Gastrointestinal Stromal Tumors
Brief Title: Imatinib Mesylate and Sunitinib in Treating Patients With Gastrointestinal Stromal Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jordan Berlin, Professor of Medicine; Clinical Director, GI Oncology Program; Director, Phase I Program; Medical Director, Clinical Trials Shared Resources; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0621; P30CA068485 (NIH); VU-VICC-GI-0621; NCT00495001 (obsolete NCT alias)
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: gastrointestinal stromal tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Drug: imatinib mesylate; Drug: sunitinib malate; Other: pharmacological study

INTERVENTIONS:
Drug: imatinib mesylate — will start at 200 mg daily and will be escalated up to 400 mg bid.If the 400 mg bid dose is tolerated, no further dose escalation will be performed. In the case of excessive toxicity on the starting dose, the option for de-escalation is provided. Sunitinib will start at 25 mg daily and if tolerated, will be escalated to 37.5 mg daily for subsequent dose levels.
  Other Names: None noted
Drug: sunitinib malate
  Other Names: none noted
Other: pharmacological study
  Other Names: Not noted

SUMMARY:
RATIONALE: Imatinib mesylate and sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of imatinib mesylate given together with sunitinib in treating patients with gastrointestinal stromal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose of imatinib mesylate in combination with sunitinib malate in patients with gastrointestinal stromal tumors.
* To determine the toxicity of this regimen in these patients.
* To determine the antitumor activity in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of imatinib mesylate.

Patients receive oral sunitinib malate once daily on days 1-14 in course 1 and on days 1-42 in all subsequent courses. Beginning in course 2, patients also receive oral imatinib mesylate once or twice daily on days 1-42. Courses repeat every 6 weeks in the absence of unacceptable toxicity.

Blood samples are collected on day 15 and day 43 for pharmacokinetics.

After completion of study treatment, patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy proven gastrointestinal stromal tumor
* Patients previously treated with imatinib mesylate must have documented progression of disease

  * Untreated disease allowed
* Must have ≥ 1 measurable lesion by RECIST
* No history of or known brain metastases, spinal cord compression,carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/μL
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 150,000/μL
* Total serum bilirubin ≤ 2.0 mg/dL
* Serum calcium ≤ 12.0 mg/dL
* Serum creatinine ≤ 1.8 mg/dL
* AST and ALT ≤ 3 times upper limit of normal (ULN) (5 times ULN if liver function abnormalities are due to underlying malignancy)
* Able to take oral medications
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No grade 3 hemorrhage within the past 4 weeks
* No myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism within the past 6 months
* No ongoing cardiac dysrhythmias ≥ grade 2
* No prolonged QTc interval on baseline EKG
* No hypertension that cannot be controlled by medications (BP > 150/100 mm Hg, despite medical therapy)
* No pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* No known HIV or AIDS-related illness or other active infection
* No other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator, preclude study entry
* No malabsorption syndrome
* No prior intolerance of imatinib mesylate or toxicity necessitating dose modification
* No prior intolerance of sunitinib malate or toxicity necessitating dose modification

PRIOR CONCURRENT THERAPY:

* Recovered from all acute toxic effects of prior chemotherapy, radiotherapy, or surgical procedures
* No major surgery or radiotherapy within the past 4 weeks
* No concurrent treatment on another clinical trial, except supportive care trials or non-treatment trials (e.g., quality of life)
* No concurrent ketoconazole and other agents known to induce CYP3A4
* No concurrent theophylline or phenobarbital and/or other agents metabolized by the cytochrome P450 system
* No ongoing therapeutic doses of coumadin, except low-dose oral coumadin up to 2 mg once daily for thrombosis prophylaxis
* No concurrent Hypericum perforatum (St. John's wort) or other herbal medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of imatinib mesylate in combination with sunitinib malate | at 6 weeks

SECONDARY OUTCOMES:
Toxicity profile as assessed by NCI CTCAE v3.0 | every 6 weeks
Pharmacokinetics | days 15 & 43
Preliminary data on anti-tumor activity of these drugs as assessed by RECIST | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jordan D. Berlin, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center; Charles D. Blanke, MD, FACP, Principal Investigator — OHSU Knight Cancer Institute; Emily Chan, MD, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee